CLINICAL TRIAL: NCT02609958
Title: A Phase 2A, Single Arm, Multicentre, Study of ASLAN001 in Patients With Advanced or Metastatic Cholangiocarcinoma Who Progressed on at Least 1 Line of Systemic Therapy
Brief Title: ASLAN001 in Patients With Advanced or Metastatic Cholangiocarcinoma Who Progressed on at Least 1 Line of Systemic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN001-005
Record Dates: First submitted 2015-11-08; First posted 2015-11-20 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — ARRY-334543

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm A (Experimental): Varlitinib (ASLAN001) tablets
  Interventions: Drug: Varlitinib

INTERVENTIONS:
Drug: Varlitinib — varlitinib tablets with:
  1. starting dose: 300mg BID
  2. target dose: 400mg BID
  3. dose modification by investigator allowed between 200mg BID to 500mg BID
  Other Names: ASLAN001; ARRY-334543; ARRY-543

SUMMARY:
This is a single arm, multicentre, Phase 2 study to assess efficacy and safety of ASLAN001 in patients with advanced or metastatic cholangiocarcinoma who progressed on at least 1 line of systemic therapy.

25 evaluable patients will be enrolled in the study. After evaluation of initial response in the first 10 evaluable patients, Sponsor will make a decision on recruitment of an additional 15 evaluable patients. If no response is observed, the study will stop.

The primary objective is to assess efficacy of varlitinib (also known as ASLAN001) as measured by ORR (based on RECIST v1.1). The secondary objectives are to (1) evaluate the efficacy of varlitinib, as measured by DoR, PFS, OS and DCR, (2) assess ORR, DoR, PFS, DCR and OS by tumor EGFR/HER2 status, (3) assess safety and tolerability of ASLAN001 monotherapy. Exploratory objectives are to explore possible relationships between response to ASLAN001 and the protein expression levels and gene mutational status of the proteins and genes via IHC and PCR/Sequencing.

DETAILED DESCRIPTION:
Cholangiocarcinoma (CCA) is a malignancy arising from the biliary epithelium characterized by poor prognosis and poor response to current treatments. Emerging at any portion of the biliary tree, it includes a group of tumours with epidemiologic, morphologic, biologic, and clinical heterogeneity. Despite recent medical advances, the long-term outcomes and recurrence rates for CCA are poor. The 5-year survival rate following surgical resection is 11-40%. Tumour recurrence rates are as high as 50-65%, with a median time to recurrence between 12-43 months.

In the United States, the incidence and mortality of CCA have increased over the last 30 years without clear underlying etiological reasons. The only curative therapy is surgical; however this is not an option for many patients given the stage of the disease at presentation and metastasis. While improvements in diagnostic modalities and neoadjuvant chemotherapy have allowed for detection at earlier stages and greater survival rates, the prognosis is still unfavorable. Therapies that can decrease tumour growth, improve resection outcomes, increase survival rates, and decrease recurrence would make a great impact on the quality of life of CCA patients and are urgently needed.

Currently, the Food and Drug Administration (FDA)-approved agents used in unresectable CCA include gemcitabine, capecitabine, cisplatin, oxaliplatin, fluoropyrimidines (including 5-fluorouracil), or a combination of these. However, none are FDA-approved primarily for use in CCA specifically. Gemcitabine and cisplatin combination therapy, along with fluoropyrimidine-based or other gemcitabine-based regimens are part of the guidelines for unresectable cancer per the National Comprehensive Cancer Network. To date, the most effective chemotherapy regimen is administration of gemcitabine with cisplatin or oxaliplatin, which have now become the standard of care for systemic therapy. Even this most efficacious treatment has been found to only modestly increase overall survival (11.7 months vs 8.3 months for patients receiving gemcitabine alone) and progression-free survival (8.4 vs 6.5 months). Standard treatment as second-line chemotherapy for CCA is unclear as there is no significant evidence for specific therapy which indicates that further chemotherapy beyond progression on first-line chemotherapy improves survival.

CCA involves mutations in members of the ErbB family, including EGFR and HER2 mutations. EGFR is overexpressed in both intrahepatic and extrahepatic CCA (30.8% and 20.9%, respectively) and is an independent prognostic factor in intrahepatic cases, per Yang et al 2014. While this study found overexpression of HER2 exclusively in extrahepatic samples (and only in 4.5% of these), previous studies have implicated this protein in both extra- and intrahepatic tumours. Settakorn et al (2005) showed HER2 expression is correlated with high histological grade in intrahepatic CCA. Kim et al. (2007) found HER2 (gene and protein levels) are overexpressed in approximately 30% of extrahepatic CCA patients and is a prognostic factor for survival in those with lymph node metastasis.

EGFR, HER2, and HER4 are single-pass transmembrane glycoprotein receptors, members of the type I receptor tyrosine kinase family. Upon ligand binding, their activation induces the homo- or heterodimerization and subsequent phosphorylation of intracellular tyrosines, which lead to both cell proliferation and survival and therefore cancer development and progression. EGFR and HER2 inhibitors have both demonstrated clinical efficacy in cancer treatment. The simultaneous inhibition of both represents a new therapeutic approach for broadly targeting different tumour types that may be more effective than selective inhibition of each receptor.

Varlitinib, also known as ASLAN001 is a potent, orally active inhibitor of the receptor tyrosine kinases epidermal growth factor (EGFR) and human epidermal growth factor receptors 2 and 4 (HER2, HER4). In cell-based assays, varlitinib has been shown to potently inhibit the phosphorylation of EGFR, HER2, and HER4 in a dose-dependent manner. In cell lines overexpressing HER2, varlitinib also inhibited the phosphorylation of the HER2 downstream effector AKT.

ASLAN hypothesises that varlitinib will inhibit EGFR, HER2, HER4 as their mutations results in CCA, thus in turn inhibiting the growth of cancerous cells and development/progression. ASLAN believes that varlitinib is a compound that may be beneficial to patients with cancer by simultaneous inhibition of these receptors.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have advanced (unresectable) or metastatic, intra or extra hepatic adenocarcinoma originated from bile duct. Histologically-confirmed diagnosis is required for the first 10 evaluable patients. The following patients could be confirmed histologically or cytologically.
* Patients must have disease progression after failing at least 1 line of systemic drug regimen for advanced cholangiocarcinoma due to disease progression or intolerance.
* Presence of radiographically measurable disease based on RECIST v1.1.
* No evidence of biliary duct obstruction, unless obstruction is controlled by local treatment or, in whom the biliary tree can be decompressed by endoscopic or percutaneous stenting with subsequent reduction in bilirubin to below 1.5 x upper level of normal (ULN).
* Patients of respective country's legal age or older at the time of written informed consent.
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patient must be able to understand and willing to sign the informed consent form and donate tumour tissue (archival or fresh) for evaluation of relevant exploratory endpoints. The first 10 evaluable patients need to have adequate archival tissues for exploratory objectives.
* Patient with adequate organ and hematological function:

  * Hematological function, as follows:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
    * Platelet count ≥ 100 x 10^9/L
  * Renal functions, as follows:

    ---Serum creatinine ≤ 1.5x ULN or eGFR > 60 mL/min/1.73m^2
  * Hepatic function, as follows:

    * Total bilirubin ≤ 1.5 x ULN
    * AST and ALT ≤ 5 x ULN

Exclusion Criteria:

* Patient with radiation or local treatment within the past 6 weeks for the target lesion(s).
* Patients with major surgical procedures within 21 days prior to study entry.
* Patient with brain lesion, known brain metastases (unless previously treated and well controlled for a period of at least 3 months).
* Patient with malabsorption syndrome, diseases significantly affecting gastrointestinal function, resection of the stomach or small bowel, or difficulty in swallowing and retaining oral medications.
* Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, diabetes, hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with any history of other malignancy unless in remission for more than 1 year. (Nonmelanoma skin carcinoma and carcinoma-in-site of uterine cervix treated with curative intent is not exclusionary).
* Female patients who are pregnant or breast feeding.
* Patients who were previously treated with Varlitinib.
* Patients who have received any investigational drug (or have used an investigational device) within the last 14 days before receiving the first dose of study medication.
* Patient with unresolved or unstable serious toxicity ( ≥ CTCAE 4.03 Grade 2) from prior administration of another investigational drug and/or prior cancer treatment.
* Patients with a known history of HIV, decompensated cirrhosis, chronic hepatitis B with HBV DNA > 2000 IU/ml or persistent abnormal ALT in the past 6 months, chronic hepatitis C with persistent abnormal ALT in the past 6 months.
* Known History of drug addiction within last 1 year.
* Patients who need continuous treatment with proton pump inhibitors during the study period.
* Any history or presence of clinically significant cardiovascular, respiratory, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease or any other condition which in the opinion of the Investigator could jeopardize the safety of the patient or the validity of the study results.

For additional information regarding investigative sites for this trial, pls contact ASLAN at contactus@aslanpharma.com

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Through study duration, estimated 3 years
  Defined as the proportion of patients with a response of PR or CR, as defined by RECIST v1.1 criteria. Data obtained up until disease progression, or last evaluable assessment in the absence of disease progression, will be included in the assessment of ORR.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Through study duration, estimated 3 years
  PFS is defined as the time from start of treatment until the date of objective disease progression or death (by any cause in the absence of disease progression) regardless of whether the patient withdraws from study therapy or receives another antitumour therapy prior to disease progression.
Disease Control Rate (DCR) | Through study duration, estimated 3 years
  Defined as proportion of patients with a best response of stable disease or better as defined by RECIST v1.1 criteria. Note, a minimum interval of 6 weeks (±5 days) from first dose is required for a patient to be attributed a best response of stable disease. Data obtained up until disease progression, or last evaluable assessment in the absence of disease progression, will be included in the assessment of DCR.
Duration of Response (DoR) | Through study duration, estimated 3 years
  Defined as the time from the date of first documented response until the date of documented disease progression or death in the absence of disease progression, the end of response should coincide with the date of disease progression or death from any cause used for the PFS endpoint. The time of the initial response will be defined as the latest of the dates contributing towards the first visit response of PR or CR.
  If a patient does not progress following a response, then their DoR will use the PFS censoring time.
Overall Survival (OS) | Through study duration, estimated 3 years
  Defined as the time from the date of start of treatment until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Safety for all advanced or metastatic Cholangiocarcinoma (CCA) subjects (Physical examination, vital signs, weight, ECG parameter, clinical laboratory tests and Adverse Events) | Through study duration, estimated 3 years
  Patient safety will be evaluated based on physical examination, vital signs (blood pressure [systolic and diastolic], resting pulse, respiratory rate, weight and body temperature), ECG parameters, clinical laboratory tests (hematology, clinical chemistry, coagulation and urinalysis) and AEs.

OTHER OUTCOMES:
Possible relationship of protein expression level and gene mutational status determined from archival material or biopsy tissue samples with response to ASLAN001. | Through study duration, estimated 3 years
  Possible relationship of protein expression level and gene mutational status determined from archival material or biopsy tissue samples with response to ASLAN001, using IHC, PCR/Sequencing and if additional material is available, IHC staining methods.

CONTACTS AND LOCATIONS:
Overall Officials: Please contact us for more information, Study Director — ASLAN Pharmaceuticals Pte Ltd
Locations (3):
- Singapore, Singapore
- Seoul, South Korea
- Taipei, Taiwan